CLINICAL TRIAL: NCT04451499
Title: The Effect of Adding Smartphone-based Platform to the Bariatric Surgery Preparation Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Medical Center (Other)
Collaborators: Ariel University (Other)
Responsible Party: Principal Investigator, Shiri Sherf Dagan, Dietitian and Epidemiologist, Assuta Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0018-20-ASMC
Record Dates: First submitted 2020-06-23; First posted 2020-06-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Bariatric Surgery Candidate; Nutritional and Metabolic Diseases
Keywords: Bariatric surgery; Nutrition; Smartphone-based education platform; Pre-surgery preparation
MeSH Terms: conditions — Nutritional and Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group -smartphone app (Experimental): All the participants will receive the standard care of 3-6 preparation to bariatric surgery meetings with a dietitian.
  All the participants will get access to our study's smartphone app site.
  Interventions: Other: Smartphone app
- Control group (No Intervention): All the participants will receive the standard care of 3-6 preparation to bariatric surgery meetings with a dietitian.

INTERVENTIONS:
Other: Smartphone app — The study specific smartphone app site will be based on current literature plus investigators experience and will include a wide knowledge on types of surgeries, dietary guidelines pre- and post-surgery, fluids type and amount, knowledge on supplementation use pre and post-surgery, general dietary knowledge, psychological information, physical activity, recommendation and tips for long-term surgery success, emphasis will be made on long-term follow-up meetings with the bariatric team and practical information on the preparation to the hospitalization process. The smartphone app site will contain video-based modules and encouraging messages. Patients will be encouraged to use the platform to ask questions and receive answers regarding any aspect of the surgery.
  Arms: Intervention group -smartphone app

SUMMARY:
A randomized controlled trial on 40 bariatric surgery candidates who will be randomized into two arms (app vs. control). All the participants will receive the standard care of 3-6 preparation to bariatric surgery meetings with a dietitian, and only those participants who will assigned to the experimental group will get access to our study's smartphone app site during this period.

Evaluations will be performed at baseline, at the end of the intervention phase (after 3-6 meetings as needed) and at 1 and 2 years post-surgery (data will be collected at 1 and 2 years post-surgery by phone calls).

Data which will be collected for this study include:demographics and medical data, anthropometrics including body composition analysis, handgrip Strength, physical activity, hydration state, bariatric surgery knowledge questionnaire, quality of life by visual analogue scale, compliance to dietary and lifestyle BS recommendations, readiness for surgery, the subject's experience regarding the smartphone app, surgical data and adherence to post-surgical follow-up by the bariatric team.

DETAILED DESCRIPTION:
A randomized controlled trial on 40 bariatric surgery candidates who will be recruited while attending to the bariatric clinics and by advertisement about the study. Patients will be randomized into two arms (app vs. control) using an online software. All the participants will receive the standard care of 3-6 preparation to bariatric surgery meetings with a dietitian, and only those participants who will be assigned to the experimental group will get access to our study's smartphone app site during this period. The study specific smartphone app site will be based on current literature plus investigators experience and will include a wide knowledge on types of surgeries, dietary guidelines pre- and post-surgery, fluids type and amount, knowledge on supplementation use pre and post-surgery, general dietary knowledge, psychological information, physical activity, recommendation and tips for long-term surgery success, emphasis will be made on long-term follow-up meetings with the bariatric team and practical information on the preparation to the hospitalization process. The smartphone app site will contain video-based modules and encouraging messages. In addition, patients will be encouraged to use the platform to ask questions and receive answers regarding any aspect of the surgery.

Evaluations will be performed at baseline, at the end of the intervention phase (after 3-6 meetings as needed) and at 1 and 2 years post-surgery (data will be collected at 1 and 2 years post-surgery by phone calls).

Data which will be collected for this study include:demographics and medical data, anthropometrics including body composition analysis, handgrip Strength, physical activity, hydration state, bariatric surgery knowledge questionnaire, quality of life by visual analogue scale, compliance to dietary and lifestyle BS recommendations, readiness for surgery, the subject's experience regarding the smartphone app, surgical data and adherence to post-surgical follow-up by the bariatric team.

ELIGIBILITY:
Inclusion Criteria:

* Pre-surgery: 18 years old or older, BMI ≥ 40 kg/m² or BMI≥35 kg/m² with comorbidities.
* Planned surgery types: LSG, RYGB and OAGB
* Reading and speaking Hebrew.

Exclusion Criteria:

* Previous bariatric surgery.
* Planned surgery types: LAGB or BPD-DS.
* Patients who underwent more than 1 preparation to bariatric surgery meeting with a dietitian.
* Patients with an active psychiatric disorder (uncontrolled) or have other contraindications to bariatric surgery such as addiction to alcohol or drugs.
* Diabetic patients taking Insulin.
* Patients who do not own a smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Changes in bariatric surgery nutrition-knowledge score | Baseline and up to 3 months (end of the intervention phase)
  Bariatric surgery nutrition-knowledge score will be measured by a validated questionnaire

SECONDARY OUTCOMES:
Changes in weight | Baseline, up to 3 months (end of the intervention phase) and 1 and 2 years post-surgery
  Weight loss
Changes in body composition | Baseline and up to 3 months (end of the intervention phase)
  Body composition will be measured using multi-frequency bioelectrical impedance analysis
Changes in functionality | Baseline and up to 3 months (end of the intervention phase)
  Handgrip muscle strength-test will be measured by a digital hand dynamometer
Changes in hydration state | Baseline and up to 3 months (end of the intervention phase)
  Patients will be asked to match the color that best describes their urine color according to a standardized urine color scale
Changes in step count | Baseline and up to 3 months (end of the intervention phase)
  Physical activity will be measured by pedometers
Changes in compliance to dietary and lifestyle bariatric surgery recommendations | Baseline, up to 3 months (end of the intervention phase) and 1 and 2 years post-surgery
  Patients will be asked if they kept the recommended behaviors by a questionnaire
Changes in quality of life: VAS scale | Baseline, up to 3 months (end of the intervention phase) and 1 and 2 years post-surgery
  Patients will be asked to rate their overall state of health from 0-100 using a VAS scale
Readiness for surgery | Up to 3 months (end of the intervention phase)
  Patients will be asked to rate their subjectively overall readiness to the surgery from 0-100 using a VAS scale
The subject's experience regarding the smartphone app | Up to 3 months (end of the intervention phase)
  Patients in the intervention arm will be ask about the ease of use
Surgical time | During surgery
  Surgery time in minutes
Adherence to post-surgical follow-up by the bariatric team | 1 and 2 years post-surgery
  Patients will be ask how many meetings they had with the bariatric team since the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No